CLINICAL TRIAL: NCT03584529
Title: Association Between Vitamin D and the Development of Uterine Fibroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2017-07-126
Record Dates: First submitted 2018-06-13; First posted 2018-07-12 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-07

CONDITIONS: Gynaecological Disease; Vitamin D Deficiency
MeSH Terms: conditions — Genital Diseases, Female; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vitamin D deficiency treatment group (Experimental): patients with vitamin D deficiency (12 ng/ml ≤ serum 25-hydroxyvitamin D3 < 20 ng/ml)and uterine fibroids receive 1600 IU/day of vitamin D3 oral capsule for two years
  Interventions: Drug: Vitamin D 3
- vitamin D deficiency control group (No Intervention): patients with vitamin D deficiency (12 ng/ml ≤ serum 25-hydroxyvitamin D3 < 20 ng/ml)and uterine fibroids receive regular follow-up.
- vitamin D insufficiency treatment group (Experimental): patients with vitamin D insufficiency (20 ng/ml ≤ serum 25-hydroxyvitamin D3 < 30 ng/ml) and uterine fibroids receive 800 IU/d of vitamin D3
  Interventions: Drug: Vitamin D 3
- vitamin D insufficiency control group (No Intervention): patients with vitamin D insufficiency (20 ng/ml ≤ serum 25-hydroxyvitamin D3 < 30 ng/ml)and uterine fibroids receive regular follow-up.

INTERVENTIONS:
Drug: Vitamin D 3 — Non-Vitamin D3 Drops group Patients in this group would take nothing.
  Arms: vitamin D deficiency treatment group; vitamin D insufficiency treatment group

SUMMARY:
the aim of this randomised clinical trial study is to evaluate whether supplementation with vitamin D could inhibit the growth of uterine fibroids in reproductive stage women.

DETAILED DESCRIPTION:
180 patients with vitamin D deficiency (12 ng/ml ≤ serum 25-hydroxyvitamin D3 < 20 ng/ml) and uterine fibroids will be randomly assigned in a ratio of 1:1 to two groups: intervention group A and control group B. 180 patients with vitamin D insufficiency (20 ng/ml ≤ serum 25-hydroxyvitamin D3 < 30 ng/ml) and uterine fibroids will be also randomly assigned in a ratio of 1:1 to two groups: intervention group C and control group D. The intervention group A will receive 1600 IU/d of vitamin D3; The intervention group C will receive 800 IU/d of vitamin D3; the control group B and the control group D will receive regular follow-up. Patients will be followed up at the same time points for 24 months. The outcome measure is the growth of uterine fibroids in different groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients are willing to cooperate with the follow-up and sign informed consent;
* 2. Females aged 35-50 who are diagnosed as having uterine fibroids by transvaginal or abdominal ultrasonography;
* 3. The maximum average diameter of intramural myoma is ≤ 4cm，≥ 1cm; The amount of myoma is less than 4;
* 4. Serum 25-hydroxyvitamin D3 < 30 ng/ml, ≥ 12 ng/ml.

Exclusion Criteria:

* 1. Patients with heavy menstrual bleeding (>80.0 mL), menstrual disorders, pelvic discomfort, infertility, or other indications for operation;
* 2. Patients complicated with myoma degeneration and adenomyosis that were suspected or diagnosed by ultrasound or gynecologic examination;
* 3. Allergic to vitamin D3;
* 4. Use of sexual hormone, mifepristone, gonadotropin-releasing hormone agonist (GnRHa), or other medication which is likely to interfere with uterine fibroids within 3 months;
* 5. Pregnancy, lactation, postmenopause, or planned pregnancy within two years;
* 6. Suspected or identified as other tumors of genital tract;
* 7. History of osteoporosis or vitamin D deficiency taking vitamin D supplements within previous one month;
* 8. History of autoimmune diseases, infectious diseases (tuberculosis, AIDS), autoimmune diseases, digestive system diseases (malabsorption, crohn disease, and dysentery);
* 9. Alanine aminotransferase (ALT) or aspartate transaminase(AST) more than 3 times of the normal upper limit, total bilirubin (TBIL) more than 2 times of the normal upper limit;
* 10. Creatinine levels≥1.4 mg/dL (123μmol/L) or creatinine clearance ≤ 50 mL/min;
* 11. History of malignant tumors;
* 12. Simultaneous participation in another clinical study with investigational medicinal product(s) or researcher thinks the subjects are not suitable for this trial.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
volume of the total fibroids | two years after treatment
  percent change in volume of the largest fibroid compared to baseline in different groups

SECONDARY OUTCOMES:
percentage of subjects undergoing other medical or surgical treatment of uterine fibroids | two years after treatment
  percentage of subjects undergoing other medical or surgical treatment of uterine fibroids
Hypercalcemia | Two years after treatment
  The level of serum calcium > 2.5 mmol/L
abnormal liver function | Two years after treatment
  Alanine aminotransferase (ALT) or aspartate transaminase (AST) more than 3 times of the normal upper limit, total bilirubin (TBIL) more than 2 times of the normal upper limit
urinary calculus | Two years after treatment
  urinary calculus
abnormal renal function | Two years after treatment
  Creatinine levels ≧ 1.4 mg/dL (123μmol/L) or creatinine clearance ≦ 50 mL/min
volume of the largest fibroid | One year after treatment
  percent change in volume of the largest fibroid compared to baseline in different groups
volume of the total fibroids | One year after treatment
  percent change in volume of the total fibroids compared to baseline in different groups
volume of the largest fibroid | two years after treatment
  percent change in volume of the largest fibroid compared to baseline in different groups

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Sheng B, Song Y, Liu Y, Jiang C, Zhu X. Association between vitamin D and uterine fibroids: a study protocol of an open-label, randomised controlled trial. BMJ Open. 2020 Nov 6;10(11):e038709. doi: 10.1136/bmjopen-2020-038709. PMID 33158822

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03584529/Prot_SAP_001.pdf